CLINICAL TRIAL: NCT06971341
Title: Retrospective Observational Study in Patients With Onychomycosis Treated With Mycoclear® and Ciclopirox
Brief Title: Study in Patients With Onychomycosis Treated With Mycoclear® and Ciclopirox
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: Dionisio Franco Barattini, MD, MBA, MSc (Unknown)
Responsible Party: Principal Investigator, Michela Valeria Rita Starace, MD PhD, Full-time Researcher RTD-B, University of Bologna
Other Study IDs: ONYCO/23
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Onychomycosis of Toenails
Keywords: onychomycosis; medical device; observational study
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mycoclear®, medical device as antimycotic topical solution: Mycoclear® was topically administered as indicated in the instructions for use of the product for a maximum of 24 weeks
- Ciclopirox, antimycotic drug: Ciclopirox was topically administered as indicated in the instructions for use of the product for a maximum of 24 weeks

SUMMARY:
The goal of this study is to learn about the effectiveness and safety of two products, ciclopirox or Mycoclear®, in treating fungal infections. People with fungal infections of the nails and over the age of 18 were treated at the Department of Dermatology, IRCCS Azienda Ospedaliero - Universitaria Sant'Orsola in Bologna (Italy) between January 1, 2019, and April 30, 2023. The people were treated as part of their regular medical care with ciclopirox or Mycoclear®. In this observational study, the data are now being reviewed to answer the following questions:

• Does Mycoclear® work as well as ciclopirox for fungal nail infections, when used for up to 24 weeks?

People were seen at the beginning for an initial assessment, and then again at two, four, 12, and 24 weeks. The doctor did the following main tests during the study period:

* Performing the clinical evaluation
* Checking the lab test for a fungal infection.
* Measuring how much of the nail grows without problems. The results of this study will help dermatologists choose the best treatment for fungal nail infections.

DETAILED DESCRIPTION:
In Italy the prevalence of onychomycosis in subjects aged >65 years was as high as 35%. This observational, retrospective study has the objective to evaluate the safety and effectiveness of two treatment for distal and lateral subungual onychomycosis (DLSO), the most prevalent clinical variant of onychomycosis. Two cohorts of patients treated between January 2019, and April 2023 are involved: 40 patients treated with Mycoclear, a medical device that is widely used as an antifungal in outpatient clinical practice and 40 patients treated with ciclopirox, an commonly used antifungal drug. The primary outcomes are the Investigator Global Assessment of Efficacy, mycological assessment, and the extent of healthy nail growth. Safety is evaluated by the incidence of adverse events. Patients were treated for a maximum period of 24 weeks, in accordance with the "standard usual care" of the center and were visited at baseline, week two, four, 12, and 24 (final visit).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients clinically and microscopically KOH diagnosed with distal and lateral subungual onychomycosis (DLSO) (≤30% involvement of the nail plate of at least one of the great toenails) and evaluated as mild to moderate following OSI6.
* Patients presenting positive direct potassium hydroxide (KOH) microscopy and positive fungal culture for dermatophytes

Exclusion Criteria:

* Other types of onychomycoses.
* Subjects who used systemic antifungal agents within 6 months or topical antifungal agents on toenails within 6 weeks of screening.
* Pregnant woman, lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal outpatients affected by distal and lateral subungual onychomycosis (DLSO) and visited in the Department of Dermatology at the IRCCS Azienda Ospedaliero-Universitaria Sant'Orsola in Bologna, Italy, between January 1, 2019, and April 30, 2023
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Investigator Global Assessment of Efficacy | 24 weeks
  Change from baseline to 24 weeks of nail color, surface, and thickness assessed by the Investigator during the medical examinations and scored by a ordinal scale as follows : 0=no change; 1=moderate improvement; 2=excellent improvement.
Mycological assessment | 24 weeks
  It was assessed by Investigator during the medical examination by KOH staining and collection of a sample for culture. It was scored according the following: negative culture=cure; positive culture=failure.

SECONDARY OUTCOMES:
Patient Global Assessment of Efficacy | 24 weeks
  Change from baseline to the final 24 week visit of global treatment effectiveness assessed by the patient and scored by a ordinal scale as follows : 0=no change; 1=moderate improvement; 2=good improvement; 3=excellent improvement.
Patient Assessment of Usability | 24 weeks
  The patient responds to a usability questionnaire for the tested medical device. The questionnaire items will be scored by an ordinal scale (ranging from 1-10) where 1 = poor rating, and 10 = excellent rating)
Incidence of adverse events | 24 weeks
  The incidence of adverse events (AEs), serious adverse events (SAEs), adverse device effects (ADEs), and serious adverse device effects (SADEs) for the two products will be collected by Investigators only if they were not reported as part of clinical practice in the previous visits performed on the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bianca M Piraccini, Prof PhD MD, Study Director — Dipartimento di Scienze Mediche e Chirurgiche Alma Mater Studiorum - Università di Bologna
Locations (1):
- UOC di Dermatologia - IRCCS Policlinico di Sant'Orsola - Università di Bologna, Bologna, BO, Italy

REFERENCES:
- [Background] Shemer A, Nathansohn N, Trau H, Amichai B, Grunwald MH. Ciclopirox nail lacquer for the treatment of onychomycosis: an open non-comparative study. J Dermatol. 2010 Feb;37(2):137-9. doi: 10.1111/j.1346-8138.2009.00773.x. PMID 20175847
- [Background] Carney C, Tosti A, Daniel R, Scher R, Rich P, DeCoster J, Elewski B. A new classification system for grading the severity of onychomycosis: Onychomycosis Severity Index. Arch Dermatol. 2011 Nov;147(11):1277-82. doi: 10.1001/archdermatol.2011.267. PMID 22106113
- [Background] Blauvelt A, Gordon KB, Lee P, Bagel J, Sofen H, Lockshin B, Soliman AM, Geng Z, Zhan T, Alperovich G, Stein Gold L. Efficacy, safety, usability, and acceptability of risankizumab 150 mg formulation administered by prefilled syringe or by an autoinjector for moderate to severe plaque psoriasis. J Dermatolog Treat. 2022 Jun;33(4):2085-2093. doi: 10.1080/09546634.2021.1914812. Epub 2021 May 5. PMID 33947295
- [Background] Yadav P, Singal A, Pandhi D, Das S. Comparative efficacy of continuous and pulse dose terbinafine regimes in toenail dermatophytosis: A randomized double-blind trial. Indian J Dermatol Venereol Leprol. 2015 Jul-Aug;81(4):363-9. doi: 10.4103/0378-6323.158634. PMID 26087080
- [Background] Arenas R. [Onychomycosis. Clinico-epidemiological mycological and therapeutic aspects]. Gac Med Mex. 1990 Mar-Apr;126(2):84-9; discussion 90-1. Spanish. PMID 2143740
- [Background] Naeimifar A, Samadi A, Ahmad Nasrollahi S, Fattahi A, Ghasemi Z, Azizzadeh-Roodpishi S, Malakooti S, Ehsani AH, Firooz A, Dowlatiy Y. Efinaconazole topical solution 10%: Formulation and efficacy assessment in the treatment of toenail onychomycosis. Mycoses. 2020 May;63(5):517-524. doi: 10.1111/myc.13062. Epub 2020 Mar 6. PMID 32048351
- [Background] Piraccini BM, Starace M, Toft A. Early Visible Improvements during K101-03 Treatment: An Open-Label Multicenter Clinical Investigation in Patients with Onychomycosis and/or Nail Psoriasis. Dermatology. 2017;233(2-3):178-183. doi: 10.1159/000478257. Epub 2017 Aug 5. PMID 28787710
- [Background] Gupta AK, Fleckman P, Baran R. Ciclopirox nail lacquer topical solution 8% in the treatment of toenail onychomycosis. J Am Acad Dermatol. 2000 Oct;43(4 Suppl):S70-80. doi: 10.1067/mjd.2000.109071. PMID 11051136
- [Background] Ricardo JW, Lipner SR. Safety of current therapies for onychomycosis. Expert Opin Drug Saf. 2020 Nov;19(11):1395-1408. doi: 10.1080/14740338.2020.1829592. Epub 2020 Oct 12. PMID 32990062
- [Background] Piraccini BM, Iorizzo M, Lencastre A, Nenoff P, Rigopoulos D. Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer: A Review of Its Use in Onychomycosis. Dermatol Ther (Heidelb). 2020 Oct;10(5):917-929. doi: 10.1007/s13555-020-00420-9. Epub 2020 Jul 23. PMID 32705532
- [Background] Piraccini BM, Starace M, Rubin AI, Di Chiacchio NG, Iorizzo M, Rigopoulos D; A working group of the European Nail Society. Onychomycosis: Recommendations for Diagnosis, Assessment of Treatment Efficacy, and Specialist Referral. The CONSONANCE Consensus Project. Dermatol Ther (Heidelb). 2022 Apr;12(4):885-898. doi: 10.1007/s13555-022-00698-x. Epub 2022 Mar 9. PMID 35262878
- [Background] Maggioni D, Cimicata A, Pratico A, Villa R, Bianchi F, Badiale SB, Piana U, Angelinetta C. Clinical Evaluation of a Topical Formulation for the Management of Onychomycosis. J Clin Aesthet Dermatol. 2020 Jul;13(7):53-57. Epub 2020 Jul 1. PMID 32983339
- [Background] Lipner SR, Scher RK. Onychomycosis: Treatment and prevention of recurrence. J Am Acad Dermatol. 2019 Apr;80(4):853-867. doi: 10.1016/j.jaad.2018.05.1260. Epub 2018 Jun 28. PMID 29959962
- [Background] Nenoff P, Reinel D, Mayser P, Abeck D, Bezold G, Bosshard PP, Brasch J, Daeschlein G, Effendy I, Ginter-Hanselmayer G, Graser Y, Hamm G, Hengge U, Hipler UC, Hoger P, Kargl A, Kolb-Maurer A, Kruger C, Malisiewicz B, Mayer J, Ott H, Paasch U, Schaller M, Uhrlass S, Zidane M. S1 Guideline onychomycosis. J Dtsch Dermatol Ges. 2023 Jun;21(6):678-692. doi: 10.1111/ddg.14988. Epub 2023 May 22. PMID 37212291
- [Background] Maskan Bermudez N, Rodriguez-Tamez G, Perez S, Tosti A. Onychomycosis: Old and New. J Fungi (Basel). 2023 May 12;9(5):559. doi: 10.3390/jof9050559. PMID 37233270
- [Background] Leung AKC, Lam JM, Leong KF, Hon KL, Barankin B, Leung AAM, Wong AHC. Onychomycosis: An Updated Review. Recent Pat Inflamm Allergy Drug Discov. 2020;14(1):32-45. doi: 10.2174/1872213X13666191026090713. PMID 31738146
- [Background] Cozzani E, Agnoletti AF, Speziari S, Schiavetti I, Zotti M, Persi A, Drago F, Parodi A. Epidemiological study of onychomycosis in older adults with onychodystrophy. Geriatr Gerontol Int. 2016 Apr;16(4):486-91. doi: 10.1111/ggi.12496. Epub 2015 May 15. PMID 25981058
- [Background] Heikkila H, Stubb S. The prevalence of onychomycosis in Finland. Br J Dermatol. 1995 Nov;133(5):699-703. doi: 10.1111/j.1365-2133.1995.tb02741.x. PMID 8555019
- [Background] Sigurgeirsson B, Baran R. The prevalence of onychomycosis in the global population: a literature study. J Eur Acad Dermatol Venereol. 2014 Nov;28(11):1480-91. doi: 10.1111/jdv.12323. Epub 2013 Nov 28. PMID 24283696